CLINICAL TRIAL: NCT00713102
Title: Surgical and Medical Emergencies on Board of European Aircraft Carriers
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Michael Sand, Dr., Ruhr University of Bochum
Other Study IDs: 004
Record Dates: First submitted 2008-07-08; First posted 2008-07-11 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Circulatory Collapse; Chest Pain; Diarrhea
Keywords: in-flight emergency
MeSH Terms: conditions — Shock; Chest Pain; Diarrhea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: The group includes 10189 patients with on board medical or surgical emergencies.

SUMMARY:
The goal of this retrospective study is to describe emergency relevant illnesses occurring in airline passengers.

DETAILED DESCRIPTION:
An epidemiologic database documenting medical and surgical emergencies across European airlines will provide access to data potentially valuable for further flight-epidemiological research. Data on medical emergencies / per rpk (revenue passenger kilometres) are sparse and often based on data from a single airline. While handling the data the regulations of the data protection act of the Ethic commission of the Ruhr-University Bochum are fully respected. As noted, evaluation of the data will be completely anonymized without any information regarding the airline or other details than the passengers illness.

Preview: The results of the study specified above will be submitted for publication in a peer review and Medline listed journal.

Study Design: Retrospective, epidemiological study for the evaluation of medical and surgical emergencies on board airliners.

Patients: In the context of a retrospective study approximately 20,000 patient data from 32 European airlines are collected and statistically evaluated.

Documentation: The direct documentation takes place through project responsible person into an electronic statistical data base.

ELIGIBILITY:
Inclusion Criteria:

* Men, women, adolescent, children and babies who have suffered from an emergency on board an European airline.

Exclusion Criteria:

* None

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men, women, adolescent, children and babies who have suffered from an emergency on board an European airline.
Sampling Method: Non-Probability Sample
Enrollment: 10189 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
All cause mortality, cause of medical or surgical emergency while on aircraft | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Benno Mann, MD, Study Chair — Department of General and Visceral Surgery, Augusta Krankenanstalt, Academic Teaching Hospital of the Ruhr-University Bochum; Michael Sand, MD, Principal Investigator — Department of General and Visceral Surgery, Augusta Krankenanstalt, Academic Teaching Hospital of the Ruhr-University Bochum, Germany
Locations (1):
- Department of General and Visceral Surgery, Augusta Krankenanstalt, Academic Teaching Hospital of the Ruhr-University Bochum, Germany, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Sand M, Bechara FG, Sand D, Mann B. Surgical and medical emergencies on board European aircraft: a retrospective study of 10189 cases. Crit Care. 2009;13(1):R3. doi: 10.1186/cc7690. Epub 2009 Jan 20. PMID 19154581